CLINICAL TRIAL: NCT01837901
Title: Transkorneale Elektrostimulation Zur Therapie Bei Retinitis Pigmentosa - Eine Prospektive, Randomisierte, Einfach Blinde Folgestudie
Brief Title: Transcorneal Electrostimulation for Therapy of Retinitis Pigmentosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okuvision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EST2
Record Dates: First submitted 2013-04-09; First posted 2013-04-23 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Retinitis Pigmentosa
Keywords: Transcorneal electrostimulation; TcES; TES
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham (Sham Comparator): OkuStim is used to determine the phosphene threshold, device is turned on but no stimulation is performed.
  Interventions: Device: Transcorneal electrostimulation
- 150% (Experimental): OkuStim is used to determine the phosphene threshold, and then to administer transcorneal electrostimulation with a stimulation strength corresponding to 150% of the patient's phosphene threshold.
  Interventions: Device: Transcorneal electrostimulation
- 200% (Experimental): OkuStim is used to determine the phosphene threshold, and then to administer transcorneal electrostimulation with a stimulation strength corresponding to 200% of the patient's phosphene threshold.
  Interventions: Device: Transcorneal electrostimulation

INTERVENTIONS:
Device: Transcorneal electrostimulation
  Other Names: OkuStim; TES; TcES

SUMMARY:
The purpose of this study is to determine the long-term effects of transcorneal electrostimulation (TcES) in patients with retinitis pigmentosa (RP). In a prior study (NCT00804102) the results of short-term stimulation showed a positive effect on the visual field and other parameters. In this study, the patients will be stimulated with either 0%, 150% or 200% of the individually determined phosphene threshold.

DETAILED DESCRIPTION:
The study was performed at the Centre for Ophthalmology, University of Tübingen, Germany. The protocol was approved by the local ethics committee. All procedures followed were in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration of 1975, as revised in 2008. Informed consent was obtained from all patients for being included in the study. The study was conducted according to the standards of GCP, the European Union Directive for Medical Devices, and the German Medical Product Law.

Patients were seen at 14 visits over a period of 78 weeks: one baseline visit (screening), followed by 12 visits (in week 1-4 weekly, then in weeks 10, 16, 22, 28, 34, 40, 46 and 52; dates varied a maximum of ± 1 week) including application of TcES for 52 weeks and one follow-up visit (in week 78, dates varied a maximum of ± 1 week).

After inclusion patients were randomly assigned to TcES with 0 mA (sham), 150% or 200% of their individual electrical phosphene threshold (EPT) current at 20 Hz.

Patients and technicians who performed kinetic perimetry, as well as full-field electrophysiology (ERG), multifocal ERG (mfERG) and dark adaptation, were blinded to the treatment group for the entire study period. The physicians who performed all other examinations and TcES were not blinded to study treatment because they were responsible for setting the stimulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject with RP (rod-cone dystrophy)
* BCVA 0.02 to 0.9
* Reliable visual field measurements
* Reliable ERG measurements
* Skillful enough to use the device at home
* Able to give consent and take part during the whole study

Exclusion Criteria:

* Diabetic retinopathy
* Neovascularisation of any origin
* After arterial or venous occlusion
* After retinal detachment
* Silicone oil tamponade
* Dry or exudative age-related macular degeneration
* Macular edema
* All forms of glaucoma
* Any form of corneal degeneration that reduces visual acuity
* Systemic diseases that are difficult to control or manage, that could endanger the normal study schedule
* Patients in a permanently poor general condition, which could hinder the regular attendance at control examinations in the clinic
* Forms of mental illness related to the bipolar affective and schizoid-affective disorders, and all forms of dementia
* Simultaneous participation in another interventional study or history of interventions whose effect may still persist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, Prof. Dr., Principal Investigator — Eberhard-Karls-Universität Tübingen
Locations (1):
- Department für Augenheilkunde, Eberhard-Karls-Universität, Tübingen, Germany

REFERENCES:
- [Background] Naycheva L, Schatz A, Rock T, Willmann G, Messias A, Bartz-Schmidt KU, Zrenner E, Gekeler F. Phosphene thresholds elicited by transcorneal electrical stimulation in healthy subjects and patients with retinal diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7440-8. doi: 10.1167/iovs.12-9612. PMID 23049087
- [Background] Gekeler F; Arbeitsgruppe Elektrostimulation des Department fur Augenheilkunde am Universitats-Klinikum Tubingen. [Transcorneal electrostimulation]. Ophthalmologe. 2012 Feb;109(2):129-35. doi: 10.1007/s00347-011-2450-6. German. PMID 22350549
- [Background] Schatz A, Rock T, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal electrical stimulation for patients with retinitis pigmentosa: a prospective, randomized, sham-controlled exploratory study. Invest Ophthalmol Vis Sci. 2011 Jun 23;52(7):4485-96. doi: 10.1167/iovs.10-6932. PMID 21467183
- [Background] Schatz A, Arango-Gonzalez B, Fischer D, Enderle H, Bolz S, Rock T, Naycheva L, Grimm C, Messias A, Zrenner E, Bartz-Schmidt KU, Willmann G, Gekeler F. Transcorneal electrical stimulation shows neuroprotective effects in retinas of light-exposed rats. Invest Ophthalmol Vis Sci. 2012 Aug 15;53(9):5552-61. doi: 10.1167/iovs.12-10037. PMID 22807300
- [Background] Rock T, Schatz A, Naycheva L, Gosheva M, Pach J, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Willmann G, Gekeler F. [Effects of transcorneal electrical stimulation in patients with Stargardt's disease]. Ophthalmologe. 2013 Jan;110(1):68-73. doi: 10.1007/s00347-012-2749-y. German. PMID 23329121
- [Result] Schatz A, Pach J, Gosheva M, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal Electrical Stimulation for Patients With Retinitis Pigmentosa: A Prospective, Randomized, Sham-Controlled Follow-up Study Over 1 Year. Invest Ophthalmol Vis Sci. 2017 Jan 1;58(1):257-269. doi: 10.1167/iovs.16-19906. PMID 28114587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the hospital's hereditary retinal degeneration clinic (Centre for Ophthalmology, University of Tuebingen, Tuebingen, Germany).
  Of 88 enrolled participants, 63 met the inclusion criteria and were randomized to treatment.
Groups:
- Sham: OkuStim was used to determine the phosphene threshold, device was turned on but no stimulation was performed.
- 150%: OkuStim was used to determine the phosphene threshold, and then to administer transcorneal electrostimulation with a stimulation strength corresponding to 150% of the patient's phosphene threshold.
- 200%: OkuStim was used to determine the phosphene threshold, and then to administer transcorneal electrostimulation with a stimulation strength corresponding to 200% of the patient's phosphene threshold.
Period: Overall Study
Arm/Group | Sham | 150% | 200%
Started | 22 | 21 | 20
Completed | 20 | 15 | 17
Not Completed | 2 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sham: Device was turned on but no stimulation was performed.
- 150%: Transcorneal electrostimulation with 150% of phosphene threshold.
- 200%: Transcorneal electrostimulation with 200% of phosphene threshold.
- Total: Total of all reporting groups
Arm/Group | Sham | 150% | 200% | Total
Number analyzed (Participants) | 20 | 15 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15) | 42 (13) | 49 (16) | 46 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 7 | 25
  Male | 9 | 8 | 10 | 27
Region of Enrollment [Number; unit: participants]
  Germany | 20 | 15 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Visual Field, III4e
Description: Change in the area measured by kinetic visual field measurement
Time Frame: one year
Measure: Mean (95% Confidence Interval); unit: deg2
Arm/Group | Sham | 150% | 200%
Number analyzed (Participants) | 20 | 14 | 17
deg2
  Baseline | 4835.29 [2723.26 to 6947.32] | 4988.43 [2799.14 to 7177.73] | 6234.59 [4226.84 to 8242.34]
  1 year | 4488.39 [2473.83 to 6502.95] | 4962.76 [2765.44 to 7160.08] | 5878.75 [3926.21 to 7831.28]

2. Primary Outcome: Visual Field, V4e
Description: Change in the area measured by kinetic visual field measurement
Time Frame: one year
Measure: Mean (95% Confidence Interval); unit: deg2
Arm/Group | Sham | 150% | 200%
Number analyzed (Participants) | 20 | 14 | 17
deg2
  Baseline | 7135.77 [4771.87 to 9499.66] | 7599.65 [5004.80 to 10194.50] | 8303.59 [6217.92 to 10389.27]
  1 year | 6730.20 [4459.71 to 9000.69] | 7641.55 [4945.26 to 10337.84] | 8112.18 [6028.01 to 10196.34]

3. Secondary Outcome: ERG B-wave
Time Frame: one year
Reporting Status: Not Posted

4. Secondary Outcome: ERG A-wave
Time Frame: one year
Reporting Status: Not Posted

5. Secondary Outcome: BCVA
Description: Best corrected visual acuity
Time Frame: one year
Reporting Status: Not Posted

6. Secondary Outcome: VFQ-25
Description: Visual Function Questionnaire (VFQ-25)
Time Frame: one year
Reporting Status: Not Posted

7. Secondary Outcome: Dark Adaptation
Description: Adaptation time, changes in pupil diameter, threshold to fullfield blue and red light is measured with a fullfield stimulus threshold test (FST) on the ESPION ERG machine (Diagnosys).
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 52 weeks treatment, follow-up visit after 72 weeks. AEs were recorded until the follow-up visit at 72 weeks.
Arm/Group | Sham | 150% | 200%
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 13/22 | 18/21 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=22) | 150% (N=21) | 200% (N=20)
Non-Ocular Adverse Events Total (General disorders) | 10 (16) | 11 (20) | 11 (17) — All AEs that were non-ocular
Macular edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Eye Symptom (Eye disorders) | 2 (2) | 14 (24) | 14 (22)
Ocular discomfort (Eye disorders) | 2 (2) | 2 (2) | 1 (4)
Ocular pain (Eye disorders) | 2 (3) | 2 (3) | 0 (0)
Subjective visual decrease (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation due to electrode (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular infection (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
General and ocular infection (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days